CLINICAL TRIAL: NCT00384397
Title: An Immunogenicity and Safety Evaluation of Two Doses of Menactra® (Meningococcal [Groups A, C, Y and W-135] Polysaccharide Diphtheria Toxoid Conjugate Vaccine) Given to Healthy Subjects at 9 and 12 Months of Age
Brief Title: A Study of 2 Doses of Menactra®, a Meningococcal Conjugate Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MTA44
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Results first posted 2011-06-02 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Meningococcal Meningitis; Measles; Mumps; Rubella; Varicella
Keywords: Menactra vaccine; Meningococcal meningitis; Measles; Mumps; Rubella; Varicella virus; Haemophilus influenzae type b; Pneumococcal conjugate vaccine
MeSH Terms: conditions — Meningitis, Meningococcal; Measles; Mumps; Rubella; Chickenpox; Haemophilus Infections | interventions — Meningococcal Vaccines; measles, mumps, rubella, varicella vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Menactra® Vaccine (Experimental): Participants will receive Menactra® vaccine at age 9 months and 12 months, respectively.
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate Vaccine
- Group 2: Menactra® + MMRV (Experimental): Participants will receive Menactra® at age 9 months followed by Menactra® and Measles-Mumps-Rubella-Varicella (MMRV) vaccines at Age 12 Months
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Group 3: Menactra® + PCV (Experimental): Participants will receive Menactra® at age 9 months followed by Menactra® and Pneumococcal Conjugate (PCV) vaccines at Age 12 Months
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Group 1: Menactra® Vaccine
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®; ProQuad®
  Arms: Group 2: Menactra® + MMRV
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®; Prevnar®
  Arms: Group 3: Menactra® + PCV

SUMMARY:
This is a Phase III, modified single-blind, randomized, parallel-group, multicenter, comparative trial in the United States designed to evaluate the immunogenicity and safety of two doses of Menactra vaccine administered alone, and concomitantly with other routine pediatric vaccines typically administered between 12 and 15 months of age.

Primary Objective:

To evaluate the antibody responses to meningococcal serogroups A, C, Y, and W-135.

Secondary Objectives:

Immunogenicity

* To evaluate the antibody responses to meningococcal serogroups A, C, Y, and W-135, when Menactra vaccine is administered alone or concomitantly with Hib and MMRV vaccines.
* To evaluate the antibody responses to meningococcal serogroups A, C, Y, and W-135, when Menactra vaccine is administered alone or concomitantly with PCV vaccine.

Safety

- To describe the safety profile within 7 and 30 days of each vaccination, and serious adverse events (SAEs) throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by medical history and physical examination.
* Aged 9 months (249 to 291 days) at the time of enrollment.
* The parent or legal guardian has signed and dated the Institutional Review Board-approved informed consent form

Exclusion Criteria:

* Serious acute or chronic disease (e.g., cardiac, renal, metabolic, rheumatologic, psychiatric, hematologic, or autoimmune disorders, diabetes, atopic conditions, congenital defects, convulsions, encephalopathy, blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic system, acute untreated tuberculosis) that could interfere with trial conduct or completion.
* Known or suspected impairment of immunologic function.
* Acute medical illness within the last 72 hours, or temperature ≥ 100.4 ºF (≥ 38.0 ºC) at the time of enrollment.
* History of documented invasive meningococcal disease or previous meningococcal vaccination.
* Known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C seropositivity as reported by the parent or legal guardian
* Received either immune globulin or other blood products within the last 3 months, or received injected or oral corticosteroids, or other immunomodulator therapy within 6 weeks of the study vaccines. Individuals on a tapering dose schedule of oral steroids lasting < 7 days and individuals (e.g., asthmatics) on a short schedule of oral steroids lasting 3 to 4 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment. Topical steroids are not included in this exclusion criterion.
* Anticipated to receive oral or injected antibiotic therapy within the 72 hours prior to the study blood draw. Topical antibiotics or antibiotic drops are not included in this exclusion criterion.
* Suspected or known hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the study vaccines or a vaccine containing the same substances. For ProQuad vaccine recipients, this includes a hypersensitivity to gelatin or a history of anaphylactic reactions to neomycin.
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular (IM) vaccination.
* Parent or legal guardian unable or unwilling to comply with the study procedures.
* Participation in another interventional clinical trial in the 30 days preceding enrollment, or participation in another clinical trial involving the investigation of a drug, vaccine, medical procedure, or medical device during the subject's trial period.
* Diagnosed with any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Received any vaccine in the 30-day period prior to receipt of study vaccine, or scheduled to receive any vaccination other than influenza vaccination and hyposensitization therapy in the 30-day period after receipt of any study vaccine. Hyposensitization therapy and influenza vaccination may be received up to two weeks before or two weeks after receiving the study vaccines. Subjects should not have received their 4th dose of Pneumococcal Conjugate (PCV) or Hib vaccine or their first dose of Measles-Mumps-Rubella-Varicella (MMRV) vaccine before enrollment.
* Personal or family history of Guillain-Barré Syndrome (GBS).
* History of seizures, including febrile seizures, or any other neurologic disorder.
* Known hypersensitivity to dry natural rubber latex (pertinent to the Menactra® vaccine needle shield)

Ages: 249 Days to 305 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1128 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (38):
- United States (38):
  - Montgomery, Alabama
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Norwich, Connecticut
  - Cocoa Beach, Florida
  - Viera, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Bardstown, Kentucky
  - Woburn, Massachusetts
  - Bridgeton, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Rochester, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Goldsboro, North Carolina
  - Laurinburg, North Carolina
  - Sylva, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Tulsa, Oklahoma
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Kingsport, Tennessee
  - Fort Worth, Texas
  - Layton, Utah
  - Ogden, Utah
  - Pleasant Grove, Utah
  - Provo, Utah
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Midlothian, Virginia
  - Norfolk, Virginia
  - Spokane, Washington
  - La Crosse, Wisconsin

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 20 September 2006 to 29 September 2007 at 71 US clinical centers.
Pre-assignment Details: A total of 1118 participants were enrolled, vaccinated, and included in data analysis.
Groups:
- Group 1: Menactra® Vaccine: Participants received one dose of Menactra® alone at age 9 months and a second dose of Menactra® at age 12 months.
- Group 2: Menactra® + MMRV: Participants received one dose of Menactra® at age 9 months and a second dose of Menactra® concomitantly with measles-mumps-rubella-varicella (MMRV) vaccine at age 12 months.
- Group 3: Menactra® + PCV: Participants received one dose of Menactra® at age 9 months and a second dose of Menactra® concomitantly with pneumococcal conjugate vaccine (PCV) at age 12 months.
Period: Overall Study
Arm/Group | Group 1: Menactra® Vaccine | Group 2: Menactra® + MMRV | Group 3: Menactra® + PCV
Started | 407 | 293 | 418
Completed | 375 | 247 | 385
Not Completed | 32 | 46 | 33
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Protocol Violation | 7 | 15 | 13
Not completed — Lost to Follow-up | 11 | 13 | 3
Not completed — Withdrawal by Subject | 14 | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Menactra® Vaccine | Group 2: Menactra® + MMRV | Group 3: Menactra® + PCV | Total
Number analyzed (Participants) | 407 | 293 | 418 | 1118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 407 | 293 | 418 | 1118
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 278.7 (10.55) | 279.8 (10.93) | 279.5 (11.11) | 279.3 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 128 | 217 | 562
  Male | 190 | 165 | 201 | 556
Region of Enrollment [Number; unit: participants]
  United States | 407 | 293 | 418 | 1118

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers ≥ 8 After Visit 2 Menactra® Vaccination as Measured by Serum Bactericidal Assay Using Human Complement (SBA-HC)
Time Frame: 30 days post-visit 2 Menactra®
Population: Antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® Vaccine | Group 2: Menactra® + MMRV | Group 3: Menactra® + PCV
Number analyzed (Participants) | 277 | 180 | 267
Percentage of Participants
  Meningococcal Serogroup A | 96 | 93 | 91
  Meningococcal Serogroup C | 100 | 99 | 98
  Meningococcal Serogroup Y | 96 | 97 | 95
  Meningococcal Serogroup W-135 | 86 | 88 | 81

2. Other Pre Specified Outcome: Percentage of Participants With Antibody Titers ≥ 4 After Visit 2 Menactra® Vaccination as Measured by Serum Bactericidal Assay Using Human Complement (SBA-HC)
Time Frame: 30 days post-Visit 2 Menactra®
Population: Antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® Vaccine | Group 2: Menactra® + MMRV | Group 3: Menactra® + PCV
Number analyzed (Participants) | 277 | 180 | 267
Percentage of Participants
  Meningococcal Serogroup A | 98 | 98 | 97
  Meningococcal Serogroup C | 100 | 100 | 99
  Meningococcal Serogroup Y | 99 | 99 | 98
  Meningococcal Serogroup W-135 | 93 | 96 | 91

3. Other Pre Specified Outcome: Meningococcal Serum Bactericidal Assay Using Human Complement Antibody Geometric Mean Titers Following Visit 2 Vaccination(s) at 12 Months.
Time Frame: 30 days post-Visit 2 Menactra®
Population: Geometric mean titers and their 95% Confidence Intervals, measured by SBA-HC, were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Menactra® Vaccine | Group 2: Menactra® + MMRV | Group 3: Menactra® + PCV
Number analyzed (Participants) | 277 | 180 | 267
Titers
  Meningococcal Serogroup A | 54.9 [46.8 to 64.5] | 52 [41.8 to 64.7] | 41 [34.6 to 48.5]
  Meningococcal Serogroup C | 141.8 [123.5 to 162.9] | 161.9 [136.3 to 192.3] | 109.5 [94.1 to 127.5]
  Meningococcal Serogroup Y | 52.4 [45.4 to 60.6] | 60.2 [50.4 to 71.7] | 39.9 [34.4 to 46.2]
  Meningococcal Serogroup W-135 | 24.3 [20.8 to 28.3] | 27.9 [22.7 to 34.3] | 17.9 [15.2 to 21]

4. Secondary Outcome: Percentage of Participants With At Least One Solicited Injection Site or Systemic Reaction Post-vaccination
Description: Injection site reactions: tenderness, erythema, and swelling at the Menactra site (Visits 1 and 2) and the measles-mumps-rubella, varicella (MMRV) and pneumococcal conjugate vaccine (PCV) sites (only Visit 2); Systemic reactions: Fever (temperature), vomiting, crying abnormal, drowsiness, appetite lost, and irritability following each vaccination.
Time Frame: 0-7 days post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® Vaccine | Group 2: Menactra® + MMRV | Group 3: Menactra® + PCV
Number analyzed (Participants) | 407 | 293 | 418
Percentage of Participants
  Any Solicited Injection Site Reaction Post-Dose 1 | 41 | 48 | 43
  Any Tenderness | 32 | 35 | 32
  Grade 3 Tenderness (Cries when limb is moved) | 1 | 0 | 0
  Any Erythema | 22 | 25 | 22
  Grade 3 Erythema (≥ 2.0 in) | 1 | 1 | 2
  Any Swelling | 11 | 15 | 11
  Grade 3 Swelling (≥ 2.0 in) | 0 | 2 | 1
  Any Solicited Injection Site Reaction Post-Dose 2 | 43 | 49 | 54
  Any Tenderness - Menactra Site | 36 | 39 | 48
  Grade 3 Tenderness (Cries when limb is moved) | 0 | 1 | 1
  Any Erythema - Menactra Site | 23 | 26 | 27
  Grade 3 Erythema (≥ 2.0 in) - Menactra Site | 1 | 2 | 3
  Any Swelling - Menactra Site | 10 | 14 | 17
  Grade 3 Swelling (≥ 2.0 in) - Menactra Site | 1 | 3 | 2
  Any Tenderness - MMRV Site | 0 | 37 | 0
  Gr 3 Tenderness (Cries when limb moved) MMRV Site | 0 | 1 | 0
  Any Erythema - MMRV Site | 0 | 23 | 0
  Grade 3 Erythema (≥ 2.0 in) - MMRV Site | 0 | 3 | 0
  Any Swelling - MMRV Site | 0 | 12 | 0
  Grade 3 Swelling (≥ 2.0 in) - MMRV Site | 0 | 2 | 0
  Any Tenderness - PCV Site | 0 | 0 | 47
  Gr 3 Tenderness (Cries when limb moved) PCV Site | 0 | 0 | 1
  Any Erythema - PCV Site | 0 | 0 | 30
  Grade 3 Erythema (≥ 2.0 in) - PCV Site | 0 | 0 | 4
  Any Swelling - PCV Site | 0 | 0 | 20
  Grade 3 Swelling (≥ 2.0 in) | 0 | 0 | 3
  Any Solicited Systemic Reaction Post-Dose 1 | 68 | 64 | 67
  Any Fever (Any Route) | 13 | 12 | 13
  Grade 3 Fever (Any Route > 103.1 ºF or > 39.5 ºC) | 1 | 2 | 2
  Any Vomiting | 16 | 14 | 15
  Grade 3 Vomiting (≥ 6 episodes per 24 hr) | 1 | 0 | 0
  Any Crying Abnormal | 34 | 36 | 33
  Grade 3 Crying Abnormal (> 3 hours) | 2 | 2 | 1
  Any Drowsiness | 31 | 30 | 30
  Grade 3 Drowsiness (Sleeps most of time) | 1 | 1 | 0
  Any Appetite Lost | 25 | 26 | 27
  Grade 3 Appetite Lost (Refuses ≥ 3 feeds/meals) | 1 | 0 | 0
  Any Irritability | 55 | 57 | 53
  Grade 3 Irritability (Inconsolable) | 2 | 2 | 2
  Any Solicited Systemic Reaction Post-Dose 2 | 64 | 74 | 68
  Any Fever (Any Route) | 16 | 26 | 22
  Grade 3 Fever (Any Route > 103.1 ºF or > 39.5 ºC) | 1 | 4 | 1
  Any Vomiting | 7 | 10 | 11
  Grade 3 Vomiting (≥ 6 episodes per 24 hr) | 1 | 1 | 0
  Any Crying Abnormal | 35 | 39 | 38
  Grade 3 Crying Abnormal (> 3 hours) | 2 | 1 | 5
  Any Drowsiness | 28 | 32 | 33
  Grade 3 Drowsiness (Sleeps most of time) | 1 | 1 | 1
  Any Appetite Lost | 26 | 32 | 32
  Grade 3 Appetite Lost (Refuses ≥ 3 feeds/meals) | 2 | 2 | 2
  Any Irritability | 52 | 61 | 57
  Grade 3 Irritability (Inconsolable) | 3 | 3 | 5

ADVERSE EVENTS:
Time Frame: Adverse events data for each participants were collected from the day of enrollment to the end of study, 9 months.
Arm/Group | Group 1: Menactra® Vaccine | Group 2: Menactra® + MMRV | Group 3: Menactra® + PCV
Serious Adverse Events (participants affected / at risk) | 16/407 | 9/293 | 17/418
Other Adverse Events (participants affected / at risk) | 210/407 | 137/293 | 222/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Menactra® Vaccine (N=407) | Group 2: Menactra® + MMRV (N=293) | Group 3: Menactra® + PCV (N=418)
Autoimmune neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Barrett's esophagus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Condyloma acuminatum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (5) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Menactra® Vaccine (N=407) | Group 2: Menactra® + MMRV (N=293) | Group 3: Menactra® + PCV (N=418)
Diarrhoea (Gastrointestinal disorders) | 38 (41) | 29 (38) | 40 (48)
Teething (Gastrointestinal disorders) | 56 (75) | 34 (54) | 43 (64)
Pyrexia (General disorders) | 32 (36) | 21 (24) | 37 (40)
Nasopharyngitis (Infections and infestations) | 29 (32) | 15 (17) | 18 (21)
Otitis media (Infections and infestations) | 69 (81) | 48 (55) | 85 (96)
Upper respiratory tract infection (Infections and infestations) | 47 (53) | 33 (37) | 81 (90)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (37) | 20 (22) | 22 (27)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 4 (4) | 13 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 33 (40) | 19 (20) | 29 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications